CLINICAL TRIAL: NCT02920879
Title: Airway Effects of PEEP During Anesthesia Induction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PC02
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Airway Management; Positive End Expiratory Pressure; Mask-ventilation; Anesthesia Induction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0 CPAP/ 0 PEEP, driving pressure 10 (Other): Patients will be preoxygenated with a CPAP-level of 0 cmH2O and after anesthesia induction, mask-ventilated with ZEEP and a driving pressure of 10 cmH2O./PEEP-level, driving pressure
  Interventions: Procedure: PEEP-level, driving pressure
- 0 CPAP/ 0 PEEP driving pressure 20 (Other): Patients will be pre-oxygenated with a CPAP-level of 0 cmH2O and after anesthesia induction, mask-ventilated with ZEEP and a driving pressure of 20 cmH2O./PEEP-level, driving pressure
  Interventions: Procedure: PEEP-level, driving pressure
- 10 CPAP / 10 PEEP, driving pressure 10 (Other): Patients will be pre-oxygenated with a CPAP-level of 10 cmH2O and after anesthesia induction, mask-ventilated with PEEP 10 cmH2O and a driving pressure of 10 cmH2O./PEEP-level, driving pressure
  Interventions: Procedure: PEEP-level, driving pressure
- 10 CPAP/ 0 PEEP, driving pressure 10 (Other): Patients will be pre-oxygenated with a CPAP-level of 10 cmH2O and after anesthesia induction, mask-ventilated with ZEEP and a driving pressure of 10 cmH2O./PEEP-level, driving pressure
  Interventions: Procedure: PEEP-level, driving pressure

INTERVENTIONS:
Procedure: PEEP-level, driving pressure — Different levels of PEEP and different levels of driving pressures during mask-ventilation at anesthesia induction.

SUMMARY:
This study investigates airway effects of PEEP during maskventilation at anesthesia induction. Four patient groups will be ventilated with different PEEP and driving pressures to evaluate time to open airway after start of positive pressure maskventilation during anesthesia induction.

DETAILED DESCRIPTION:
The use of continuous positive pressure (CPAP/PEEP) during pre-oxygenation and mask-ventilation in patients undergoing anesthesia induction is increasing. Continuous positive pressures have several respiratory benefits with well-documented data on both spontaneously breathing patients and intubated patients. However the effects of PEEP on anesthetized patients during mask-ventilation is poorly investigated. In a previous trial the that the investigators conducted, a PEEP-level of 10 cmH2O during mask ventilation after anesthesia induction surprisingly delayed time to alveolar ventilation compared to ZEEP. In order to investigate this phenomenon, four groups of patients will be compared during preoxygenation and mask ventilation after anesthesia induction.

Each group consisting of 30 patients will be pre-oxygenated and mask ventilated with different CPAP/PEEP levels and different driving pressures. Time to open airway is measured as number of respiratory cycles until detection of CO2 on the capnograph.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18- ≤ 65 years male or female.
2. Elective surgery under general anesthesia
3. ASA-classification 1-3
4. Signed and dated informed consent

Exclusion Criteria:

1. BMI > 30
2. Predicted difficult mask-ventilation
3. Known hiatus hernia or GERD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Time to open airway | 20 minutes
  Time to open airway depending on ventilatory settings